CLINICAL TRIAL: NCT05175703
Title: A Prospective, Multi-centre, Sinlge Arm, Post-market Registry to Assess the Clinical Performance and Safety of the Passeo-18 Lux Paclitaxel Releasing Balloon Catheter in Infrainguinal Arteries
Brief Title: Post-market Registry to Assess the Clinical Performance and Safety of the Passeo-18 Lux in Infrainguinal Arteries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Je Hwan Won, Professor, Ajou University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AJIRB-DEV-DE4-17-478
Record Dates: First submitted 2021-10-26; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Angioplasty, Balloon; Disease, Peripheral Artery
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: The Passeo-18 Lux DCB
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- the infrainguinal arteries disease group (Other): Actual patient group with any atherosclerotic change in the infrainguinal arteries
  Interventions: Device: Passeo-18 Lux Paclitaxel releasing Balloon Catheter

INTERVENTIONS:
Device: Passeo-18 Lux Paclitaxel releasing Balloon Catheter — collect short term and long term clinical evaluation data of the Passeo-18 Lux Paclitaxel releasing balloon catheter, subject to patients who visit hospital from arteriosclerosis in the infrainguinal arteries in actual clinical environment.

SUMMARY:
The purpose of his study is to collect short term and long term clinical evaluation data of the Passeo-18 Lux Paclitaxel releasing balloon catheter, subject to patients who visit hospital from arteriosclerosis in the infrainguinal arteries in actual clinical environment.

Research institute for enrollment, and period; It is planned to enroll about 200 subjects in 9 domestic research institutes. It is expected to require about 12-18 months to enroll the subjects.

Subject follow-up schedule; Perform follow-up by phone call or clinical assessment at 1, 6, 12, and 24 months of the postoperative time point

DETAILED DESCRIPTION:
This study is a prospective, multicenter, single arm, post-market registry subject to all the patient group with the relevant indications, where follow-up is performed in 1, 6, 12 (including angio follow up), and 24 month. The Passeo-18 Lux DCB including all the target patient group, is subject to every disease requiring revascularization in the infrainguinal arteries and is going to use the Passeo-18 Lux DCB.

The subject will receive percutaneous intervention using Passeo-18 Lux DCB according to the standard care guideline of this hospital. All complications and adverse events occurring during the operation will be recorded thoroughly. During the intervention, the number of lesions to be treated with Passeo-18 Lux will be determined carefully under judgment of the PI (When using more than one Passeo-18 Lux in a patient, maximum drug release recommended in the IFU should be considered.) The target lesion which is compose of one or several small lesions treatable with a balloon catheter is defined as a "treatment segment". The results of all the lesions treated with Passeo-18 Lux for the first time (regardless of which side limb) are going to be documented in eCRF, through which final results will be analyzed. All complications and adverse events from the intervention will be recorded thoroughly and reported to IRB according to the prescribed form.

Stent insertion into the lesion finishing treatment with drug coated balloon catheter will be determined by the study physician. For the subjects follow-up via phone call or clinical assessment will be conducted under below schedule. In this study the subjects who require stent insertion will not be classified as treatment failure. Before discharge of the subjects, medical prescription will follow the standard of care of this hospital, which will be documented. All the postoperative complications and adverse events will be recorded thoroughly and reported to IRB via suitable form. The subjects will be administered with proper anticoagulant, antiplatelet drug, and blood vessel dilator according to common and standard care guideline. The treatment follows the guideline described in IFU of Passeo-18 Lux DCB.

A subject does not have to participate in this study for treatment of the stenosed lower limb blood vessel. For example, there are a lot of devices available for treatment of the subject, including standard drug coated balloon, laser, and stent. The study physician will provide sufficient explanation on these alternative therapies for his/her understanding. Even though a subject decided not to participate in this study, it would not affect current and future treatment that he/she receives.

As the subjects of this study participate in in this study voluntarily according to their own will, they can discontinue the participation without any disadvantage or limitation at any time when they desire. They will not receive any disadvantage in later treatment from that. However the information collected during participation may be able to be used as it was anonymized. When a subject discontinued participation of study early, the participation should be terminated after completing preparation of eCRF as soon as possible. Also, The principal investigator regards a case as failure in follow-up of a subject up to for 24 months. In failing the follow-up, the principal investigator should record the failure of follow-up on the CRF.

ELIGIBILITY:
Inclusion Criteria:

* Person over 19 years old who is recognized as an adult in the civil law
* Person willing to sign a subject written consent
* Patient having infrainguinal arterial lesion that is adequate to intravascular treatment using Passeo-18 Lux Paclitaxel releasing Balloon Catheter
* Peripheral arterial disease in 2-5 grade of Rutherford
* Patient without at least one of significant lesions (≥50% of stenosis) in distal leaking artery. When there is at least one of opening blood vessels under the knee in treatment of arterial popliteal or at least one of opening cural vessel under the ankle in arterial treatment under the knee. Treatment of inflow arterial disease is allowed before the relevant treatment.)

Exclusion Criteria:

* Life expectancy ≤ 1 year
* Patient who is currently under medication of an investigation drug or treatment by a device that did not reach the primary endpoints.
* Subject during pregnancy or having a plan of pregnancy during the study period
* A guide wire could not passed into the target lesion (Successful passage of guide wire means its movement into the distal part of target lesion without causing arterial dissection or perforation by the end of guidewire.)
* Acute thrombosis is accompanied
* Major amputation is planned There is medical history of bypass surgery on target vessel

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinical primary endpoints | 30 days
  No occurrence of Major Adverse Event (MAE); No death or lower limb amputation in the subject from the index procedure for 30 days
Clinical primary endpoints | 6 months
  No occurrence of Major Adverse Event (MAE); No target vessel revascularization (TVR) within 6 months from index procedure.
Functional primary endpoints | 12 months
  No target lesion revascularization (TLR) (a case showing at least 50% stenosis in visual inspection of target vessel in the patient with any recurred symptom) is needed clinically for 12 months after operation.

SECONDARY OUTCOMES:
TLR (Target Lesion Revascularzation) rate | 6-24 months
  ratio of TLR patients among full cohort within 6 ~ 24 months
TVR rate | 6-24 months
  ratio of TVR patients among full cohort within 6 ~ 24 months
Survival without amputation | 6-24 months
  Survival without amputation (survival without whole amputation including minor and major amputation) for 6, 12, and 24 months after operation
device success | during index procedure
  definition of device success : Successful guide, inflation, deflation, and withdrawal of the Passeo-18 Lux Paclitaxel releasing balloon catheter
Technical success | during index procedure
  definition of technical success : Finished vascular procedure successfully and achieved ≤50% residual stenosis rate when assessing under visual inspection immediately after operation
Success in operation | during index procedure
  definition of op : Defined it as the case that technical success and device success were achieved and no MAE occurred during the index procedure period.

CONTACTS AND LOCATIONS:
Overall Officials: Je Hwan Won, MD, Principal Investigator — Korean Society of Interventional Radiology
Locations (1):
- Ajou University Hospital, Suwon, Kyunggi, South Korea

IPD SHARING:
Plan to Share IPD: No